## VALIDITY AND RELIABILITY OF REBEE WEARABLE SENSOR TO MEASURE KNEE JOINT RANGE OF MOTION

BY Ahmed Mohamed Ahmed Saleh B.Sc.in Physical Therapy, 2014

A protocol submitted in partial fulfillment of the requirements for the master degree in physical therapy for basic science Faculty of Physical Therapy

Cairo University

November 10, 2020

## **Supervisors**

Prof. Dr. Wadida Hassan Professor of Physical Therapy Basic Science Department Faculty of Physical Therapy Cairo University

Dr. Rania Reda Mohamed Lecturer of Physical Therapy Basic Science Department Faculty of Physical Therapy Cairo University

## **Contents**

| LIST OF ABBREVIATIONS | 4 |
|---------------------------------------|-----|
| CHAPTER I | |
| INTRODUCTION | |
| Introduction | 5 |
| Statement of the Problem | |
| Purpose of the Study | |
| Significance of the Study | 6 |
| Hypotheses | 7 |
| Basic Assumption | |
| Delimitations | 8 |
| CHAPTER II | |
| LITERATURE REVIEW | |
| Range of Motion | 9 |
| Causes of ROM Limitation | 9 |
| Physical Examination of ROM | 10 |
| Universal Goniometer | 10 |
| Inclinometer | 10 |
| Digital Goniometer | 12 |
| Rebee Wearable Sensor | 13 |
| CHAPTER III | |
| SUBJECTS, MATERIALS AND METHODS | |
| Design of the Study | 14 |
| Participants | 14 |
| Selection of Subjects | .14 |
| Inclusion Criteria | .14 |
| Instrumentation | .15 |
| Procedure for testing Validity | |
| Procedure for testing Reliability | |
| Knee Active ROM Measurement | |
| Steps for Using Rebee Wearable Sensor | |
| Statistical Analysis | |
| Ethical Considerations. | |
| REFERENCES | 23 |
| APPENDIX | |
| Appendix I: Patient Consent Form | 26 |

## **LIST OF ABBREVIATIONS**

APPS : Applications

AROM: Active Range of Motion

BMI : Body Mass Index

ROM: Range OF Motion

UG : Universal Goniometer

# CHAPTER I INTRODUCTION

Range of motion (ROM) of the joint is one of the factors that determine function of the musculoskeletal system. This parameter should be measured and recorded by a valid and reliable method (Yaikwawongs et al., 2009). It is considered to be an essential component of lower limb physical examination, which can be applied using various instruments such as goniometers and inclinometers (Pourahmadi et al., 2017).

Range of motion of the knee joint is one of the major factors determining the outcome after knee injuries. It is also an important measurement required by many knee scoring systems to determine the preoperative status and postoperative outcome (Anouchi et al., 1996). Measurements are used by physical therapists to quantify limitations of motion, used to decide an appropriate therapeutic interventions, and document the effectiveness of these interventions. The ideal measuring device should give reproducible valid and reliable data (Yaikwawongs et al., 2009).

Two-arm digital goniometer is still widely used in measuring uniaxial ROM of joint of extremity, there is high validity, intra rater and interrater reliability of the digital goniometer. It is considered valid and reliable tool that simplify physical therapists' work (Svensson et al., 2019).

The measurement of joint ROM is required an essential skill in the musculoskeletal assessments commonly performed by physiotherapists. The digital goniometer is the most commonly utilized clinical tool for measuring joint range of motion, the evolution of sensors technology and applications are easy to use, relatively inexpensive, and highly accessible (**Keogh et al., 2019**).

Rebee is a wearable motion sensor package of sensor with its own mobile application, which measures range of joint movement in different planes easily which the patient able to wear the sensor and move easily to measure ROM and record the measurement at the application software, that is facilitate the tele-measurement which the patients are supposed to put on the sensors and perform the actions themselves, or with assistance from physical therapist.

So this study will be conducted to test the criterion related validity and intrarater reliability of the rebee wearable sensor in measuring active knee joint ROM compared with digital goniometer measurement.

#### **Statement of the Problem**

- 1- Is the rebee wearable sensor valid to measure active knee joint ROM compared with digital goniometer measurement?
- 2- Is the rebee wearable sensor reliable in measuring active knee joint ROM?

#### **Purpose of the Study**

Purpose of the study to test the criterion related validity and intrarater reliability of rebee wearable sensor in measuring active knee joint ROM compared with digital goniometer measurement.

### **Significance of the Study**

Measurement the joint ROM with the digital goniometer is considered time consuming and difficult with respect to repeated measurements. (Svensson et al., 2019).

So there is a need to the sensors system which could be considered as a clinical measurement for ROM which will reflect in rehabilitation process through measuring the patient ROM easily (Hamel et al., 2008).

Some researchers would prefer taking the ROM of lower limb in a more functional way such as standing and walking given that the sensors were developed, which the patients are supposed to put on the sensors where the sensor placed on prominent bony landmarks at the level of lateral malleolus. It will be stabilized on the testing limbs by elastic bands and perform the actions themselves, with or without the supervision from the physical therapist (Vohralik et al., 2015).

With the use of rebee wearable sensor, the ROM of knee joint flexion and extension can be monitored easily and recorded, that lead to facilitation of tele rehabilitation. Which the patients are supposed to put on the sensors and perform knee flexion and extension themselves, with or without the supervision from the clinicians.

#### **Hypotheses**

It is hypothesized that:

- 1. Rebee wearable sensor will not be valid to measure active knee joint flexion ROM compared with digital goniometer measurement.
- 2. Rebee wearable sensor will not be valid to measure active knee joint extension ROM compared with digital goniometer measurement.
- 3. Rebee wearable sensor is not reliable to measure active knee joint flexion ROM.
- 4. Rebee wearable sensor is not reliable to measure active knee joint extension ROM.

#### **Basic Assumption**

It is assumed that:

- The movement applied will be the same for all participants and will be the same for each participant repeatedly.
- All participants will comply with the instructions honestly.
- All participants will have the same psychophysiological condition during the treatment period.

#### **Delimitations**

#### The principles respected in selecting the cases and data recording are:

- 1- 40 normal participant will be assigned to group, this number detected by G\*power 3.1 software (Universities, Dusseldorf, Germany) was used for calculation.
- 2- The participant's age ranged from 35 to 45 (Miranda et al., 2002).
- 3- The participant from both sex (Correll et al., 2018).
- 4- Participant Body mass index (BMI) from (19 to 25) normal weight (Weisell et al., 2002).
- 5- Knee flexion and extension ROM will be measured with the digital goniometer.
- 6- Knee flexion and extension ROM will be measured with the rebee wearable sensor.
- 7- The procedures will repeated two times with one week interval between measurements.

## CHAPTER II LITERATURE REVIEW

#### Range of Motion

Range of motion of the joint is the arc of motion that occurs at a joint, it is one of the factors that determine function of the musculoskeletal system. This parameter should be measured and recorded by a reproducible only method (Yaikwawongs et al., 2009)

The assessment of joint range of motion (ROM) is an important component of a physical therapy examination. These measurements are critical for providing baseline data, determining functional limitations, and monitoring changes in joint mobility in response to treatment. Measurement of ROM may also be used to detect asymmetry and movement restrictions that may increase risk of injury (Clarkson et al., 2005).

Range of motion of the knee joint is one of the major factors determining the outcome after knee injuries. It is also an important measurement required by many knee scoring systems to determine the preoperative status and postoperative outcome (Anouchi et al., 1996).

#### **Causes of ROM Limitation**

Reduced range of movement is where there is a limitation of movement at a joint. Types of reduced range of movements are:

- Muscle Injury
- Ligament injury
- Pain
- Swelling
- Arthritis (Konor et al., 2012)

#### **Physical Examination of ROM**

Each specific joint has a normal range of motion that is expressed in degrees. The reference values for the normal ROM in individuals differ slightly depending on age and gender. For example, as an individual ages, they typically lose a small amount of ROM (Yaikwawongs et al., 2009).

Analog and traditional devices to measure range of motion in the joints of the body include the goniometer and inclinometer which use a stationary arm, protractor, fulcrum, and movement arm to measure angle from axis of the joint.

Over the years, the most common instrument used for joint measurement in physio-therapy has been the universal goniometer (UG) (Norkin et al., 1995). Important psychometric characteristics of this instrument, such as intratester and intertester reliability, have been examined in many research studies. In the clinical setting, these characteristics are important because patients are often treated and reassessed, either by the same or by different physical therapists (Gogia et al., 1987).

Many research studies have found the UG to have overall good intratester and intertester reliability. However, the majority of these studies have found intratester reliability to be greater than intertester reliability (Roach et al., 1991)



In addition to the goniometer, another device being used by some clinicians to measure range of motion is the digital inclinometer. The inclinometer is similar to the goniometer in that both are lightweight and portable. However, the inclinometer has significantly more associated cost. The inclinometer has been demonstrated to possess good to excellent reliability and concurrent validity with the universal goniometer (Clarkson et al., 2005)



The digital goniometer is the most commonly utilized clinical tool for measuring joint range of motion, it gives the physiotherapist a useful method to diagnose musculoskeletal function in terms of ROM, monitor the progress of an intervention (Yaikwawongs et al., 2009).



There is high validity, intra rater and interrater reliability of the digital goniometer (Svensson et al., 2019).

To measure joints with the digital goniometer is considered time consuming and difficult with respect to repeated measurements. (Svensson et al., 2019), so there is a need to a new device that sensors system could be considered as a clinical measurement for ROM which will reflect in rehabilitation process (Hamel et al., 2008).

New evolution for measuring ROM called rebee wearable sensor. With the use of rebee wearable sensor, the ROM of knee joint flexion and extension can be monitored easily, that lead to facilitation of tele rehabilitation. Which the patients are supposed to put on the sensors and perform knee flexion and extension themselves, with or without the supervision from the clinicians.



The patients are supposed to put on the sensors and perform the actions themselves, with or without the supervision from the clinicians/ research. The evolution of sensors technology and applications are easy to use, relatively inexpensive, and highly accessible (**Keogh et al., 2019**)

# CHAPTER III SUBJECTS, MATERIALS AND METHODS

This study will be conducted at the Outpatient Clinic of Faculty of Physical Therapy, Pharos University, Alexandria, Egypt. to test the criterion related validity and reliability of rebee wearable sensor in measuring Active Knee Joint ROM compared with digital goniometer measurement.

#### **Design of the Study**

The study is Cross Section Study (Observational study).

#### **Participants**

40 normal participant will be assigned to one group, this number detected by G\*power 3.1 software (Universities, Dusseldorf, Germany) was used for calculation.

#### **Selection of Subjects**

The participant will be recruited from faculty, staff, and students of Pharos University, Egypt. Graduate Program in Physical Therapy after achieving the inclusion and exclusion criteria. Each participant will sign an informed consent before beginning of the study to insure complete satisfaction (Appendix 1)

#### **Inclusion Criteria**

- 1. 40 normal participant's age ranged from 35 to 45. (Miranda et al., 2002)
- 2. The participant from both sex. (Correll et al., 2018)
- 3. Participant Body mass index (BMI) from (19 to 25) normal weight (BMI= weight (kg) / [height (m)]<sup>2</sup>) (Weisell et al., 2002).

#### **Instrumentations**

1. Digital goniometer.

The digital goniometer will be used as a valid and reliable ROM measurement tool, the type of digital goniometer will be used in the study called digital absolute axis goniometer with accuracy about 0.99(Correll et al., 2018)

2. Rebee wearable sensor and application by XCLR8 Technologies.

The package of sensor and application will be used for measure, interpret and store participant measurement for test the criterion related validity and intrarater reliability of rebee wearable sensor in measuring active knee joint ROM

3. Health weight scale for weight and height measurement to calculate BMI. (BMI= weight (kg) / [height (m)]<sup>2</sup>) (Weisell et al., 2002).

#### **Procedure for testing Validity**

The digital goniometer will be used as a valid and reliable ROM measurement tool to be compared with rebee wearable sensor in measuring active knee joint ROM.

#### **Measure AROM of Knee Flexion with Digital Goniometer**

The participant will be at supine position with the testing knee extended, which allows assessment of the joint ROM without interference from tightness in the rectus femoris muscle, axis location at lateral epicondyle of the femur, stationary arm will be along the femur to the greater trochanter, The movement arm will be along the fibula to lateral malleolus.

The participant will asked to flex the testing knee fully through available ROM and the therapist will record the measurement to compare with rebee wearable sensor measurement.

#### Measure AROM of Knee Extension with Digital Goniometer

The participant will be at supine position with the testing knee flexed, which allows assessment of the joint ROM without interference from tightness in the rectus femoris muscle, axis location at lateral epicondyle of the femur, stationary arm will be along the femur to the greater trochanter, The movement arm will be along the fibula to lateral malleolus.

The participant will asked to extent the testing knee fully through available ROM and the therapist will record the measurement to compare with rebee wearable sensor measurement.

The following picture illustrate that measurement with the digital goniometer will be from the similar supine position of measurement with the conventional goniomtere



#### **Procedure for testing Reliability**

Designed according to Guidelines for reporting Reliability and Studies, investigating the intrarater reliability of a rebee wearable sensor will be conducted. The study will be designed in accordance with the ethical guidelines from the Helsinki declaration of ethical principles (World Medical Association (Kottner et al., 2011)).

Written consent will be retrieved from all subjects before participating in the study, the procedures will repeated two times with one week interval between measurements. Researcher will records all the measurement.

#### **Knee Active ROM Measurement with Rebee Wearable Sensor**

This process postulated by Kimberlin, 2008

To detect the joints ROM, the sensors were placed in the most distal part of the limbs with prominent bony landmarks at the level of lateral malleolus. It will be stabilized on the testing limbs by elastic bands. With the sensor light facing Lateral malleolus

#### Measure AROM of Knee Flexion with Rebee Wearable Sensor

The participant will be standing in upright position, the sensor position at the level of the Lateral malleolus, participant will be asked to flex the testing knee fully while standing supported in one leg.

#### Measure AROM of Knee Extension with Rebee Wearable Sensor

The participant will sitting at the edge of plinth with knee flexed, the sensor position at the level of the Lateral malleolus, participant will be asked to extent the testing knee through the full ROM.



The Digital goniometer and rebee wearable sensor will be used for comparison of their validity for measuring knee joint flexion and extension ROM.

Rebee wearable sensor will be used as mentioned above and this procedures will repeated two times with one week interval between measurements to test its reliability. Researcher will records all the measurement.

#### **Steps for Using Rebee Sensor Package**

1- Take the charging end of the charging cable and look for the charging port on the sensor.



2- Making sure the cable aligns with the port then connect the charger.



- 3- The USB end of the charging cable must be connected to a USB port / USB charger.
- 4- Check the sensor for a red LED light to know that it is successfully charging. The red LED will turn off once the device is fully charged.



5- Wearing the devise at the level of the Lateral malleolus with the sensor light facing Lateral malleolus.



6- Connecting the sensor to the device



Step a: Switch on the sensor device.

Step b: Go to phone's settings and turn on device's Bluetooth.

7- Look for "HC-06" (Default sensor name) under "Available devices" and tap on it.



8- Identifying the Sensors to Software



Step a: Connect the sensor you are trying to identify Step b: Look for the sensor in the list with the name "HC-06"

#### **Statistical Analysis**

Statistical methods will be used to calculate the reliability and validity of our measurements will be descriptive statistics for mean and standard deviation, also the Pearson product-moment correlation coefficient (r), an assessment of covariance.

#### **Ethical Considerations**

- 1. All participant will sign a consent form to declare that they are not forced to participate in this study. (Appendix I)
- 2. The study will be conducted after approval of ethical committee of the Faculty of physical therapy, Cairo University, Egypt.

#### **REFERENCES**

Pourahmadi, M. R., Ebrahimi Takamjani, I., Sarrafzadeh, J., Bahramian, M., Mohseni-Bandpei, M. A., Rajabzadeh, F., & Taghipour, M. (2017). Reliability and concurrent validity of a new iphone goniometric application for measuring active wrist range of motion: a cross-sectional study in asymptomatic subjects. Journal of anatomy, 230(3), 484-495.

Keogh, J. W., Cox, A., Anderson, S., Liew, B., Olsen, A., Schram, B., & Furness, J. (2019). Reliability and validity of clinically accessible smartphone applications to measure joint range of motion: A systematic review. PloS one, 14(5), e0215806.

Dobkin, B. H. (2013). Wearable motion sensors to continuously measure real-world physical activities. Current opinion in neurology, 26(6), 602.

Lewis, E., Fors, L., & Tharion, W. J. (2010). Interrater and intrarater reliability of finger goniometric measurements. American Journal of Occupational Therapy, 64(4), 555-561.

Hamel, M., Fontaine, R., & Boissy, P. (2008). In-home tele-rehabilitation for geriatric patients. IEEE Engineering in Medicine and Biology Magazine, 27(4), 29-37.

Vohralik, S. L., Bowen, A. R., Burns, J., Hiller, C. E., & Nightingale, E. J. (2015). Reliability and validity of a smartphone app to measure joint range. American journal of physical medicine & rehabilitation, 94(4), 325-330.

Correll, S., Field, J., Hutchinson, H., Mickevicius, G., Fitzsimmons, A., & Smoot, B. (2018). Reliability and validity of the halo digital goniometer for shoulder range of motion in healthy subjects. International journal of sports physical therapy, 13(4), 707.

Svensson, M., Lind, V., & Löfgren Harringe, M. (2019). Measurement of knee joint range of motion with a digital goniometer: A reliability study. Physiotherapy Research International, 24(2), e1765.

Miranda, H., Viikari-Juntura, E., Martikainen, R., & Riihimäki, H. (2002). A prospective study on knee pain and its risk factors. Osteoarthritis and cartilage, 10(8), 623-630.

Yaikwawongs, N., Limpaphayom, N., & Wilairatana, V. (2009). Reliability of digital compass goniometer in knee joint range of motion measurement. Medical journal of the Medical Association of Thailand, 92(4), 517.

Mohammadbeigi, A., Mohammadsalehi, N., & Aligol, M. (2015). Validity and reliability of the instruments and types of measurements in health applied researches. Journal of rafsanjan university of medical sciences, 13(12), 1153-1170.

Kimberlin, C. L., & Winterstein, A. G. (2008). Validity and reliability of measurement instruments used in research. American journal of health-system pharmacy, 65(23), 2276-2284.

Anouchi, Y. S., McShane, M., Kelly Jr, F., Elting, J., & Stiehl, J. (1996). Range of motion in total knee replacement. Clinical Orthopedics and Related Research (1976-2007), 331, 87-92.

Norkin CC, White DJ. (2003) Measurement of Joint Motion, a Guide to Goniometry. 3rd ed. Philadelphia: FA Davis;

Clarkson HM. (2005) Joint Motion and Function Assessment: A Research Based Practical Guide. Philadelphia, PA: Lippincott Williams & Wilkins;

Konor MM, Morton S, Eckerson JM, et al (2012): Reliability of three measures of ankle dorsiflexion range of motion. Int J Sports Phys Ther; 7:279Y87

Norkin, C. C., & White, D. J. (1995) Measurement of joint motion: a guide to goniometry... Philadelphia: FA Davis.

Roach, Kathryn E., and Toni P. Miles. (1991) "Normal hip and knee active range of motion: the relationship to age." Physical therapy 71.9: 656-665.

Clarkson, H. M. (2005). Joint motion and function assessment: a research-based practical guide. Lippincott Williams & Wilkins.

Weisell, R. C. (2002). Body mass index as an indicator of obesity. Asia Pacific journal of clinical nutrition, 11, S681-S684.

## Appendix I Patient Consent Form

I am freely and voluntarily consent in this research study under the direction of the researcher /Ahmed Mohamed Ahmed Saleh. A thorough description of the procedure has been explained to me and I understand that I can withdraw my consent and discontinue participation in this research at any time without prejudice to me.

| Participant: | Signature: |
|--------------|------------|
| Researcher: | Signature: |
| Date: | |